CLINICAL TRIAL: NCT00777049
Title: A Phase II, Open-label Multicenter Trial of Panobinostat Monotherapy in Women With HER2-negative Locally Recurrent or Metastatic Breast Cancer
Brief Title: Study of Panobinostat Monotherapy in Women With HER2-negative Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Research in Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIO 017
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ER+ and/or PgR+ (Arm I) (Experimental): Panobinostat oral 40 mg (3 times a week) given every other week as part of a 28 day cycle.
  Interventions: Drug: Panobinostat
- ER- and PgR- (Arm II) (Experimental): Panobinostat oral 40 mg (3 times a week) given every other week as part of a 28 day cycle.
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Hard gelatine capsule - 5mg and 20mg
  Other Names: LBH589

SUMMARY:
The purpose of the study is to assess the benefit of oral panobinostat monotherapy given to women with HER2-negative locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
This was a phase II, open label, multi-centre, two-arm, two-stage design, international study of oral panobinostat in women with HER2-negative locally recurrent or metastatic breast cancer.

In the first stage of the trial, 21 evaluable patients HR+ (ER+ and/or PgR+), HER2-negative, were to be treated (Arm I); if less than 3 responses were observed, that arm would be stopped and the treatment in this patient population would be declared as ineffective. In the other arm, 27 evaluable patients HR- (ER- and PgR-), HER2-negative, were to be treated (Arm II); if less than 2 responses were observed, that arm would be stopped and the treatment in this patient population would be declared as ineffective.

Given these protocol conditions, the study was stopped in Arm II due to low recruitment as there was insufficient data available to draw conclusions regarding efficacy in that arm. It should also be noted that only one response was observed in this group.. In Arm I, among the 25 evaluable patients, the study did not achieve the required number of tumor responses to allow enrolment to continue.

As such the protocol was amended to stop enrolment and remove analysis of the initially planned secondary objectives (Progression Free Survival and Overall Survival) considering the small study sample size. The patients already included were given the option to continue in the study until they reached their planned end-of-study visit.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study-related procedures
* Women ≥ 18 years old
* Patients with an ECOG performance status of ≤ 2 assessed within 2 weeks (14 days) prior to registration
* Histologically or cytologically confirmed breast cancer with locally recurrent or radiological evidence of metastatic disease. Locally recurrent disease must not be amenable to resection with curative intent.
* Measurable disease per RECIST (Response Evaluation Criteria in Solid Tumor) guidelines
* HER2-negative patients by local laboratory testing (IHC 0 or 1+ staining, IHC 2+ staining but in situ hybridization negative, or in situ hybridization negative).
* ER and PgR testing from a local laboratory is required prior to patient registration
* For Arm I: at least two lines of prior endocrine therapy (in adjuvant and/or metastatic settings) are required. Up to two prior cytotoxic chemotherapies are allowed in the metastatic setting (prior adjuvant and neoadjuvant chemotherapy is allowed).
* For Arm II: up to 2 prior cytotoxic chemotherapy regimens for treatment of metastatic or locally recurrent breast cancer are allowed.
* Complete radiological tumor measurement within 4 weeks (28 days) prior to registration:

  * Chest: CT scan with intravenous contrast if the contrast is not medically contraindicated or MRI
  * Abdomen: CT scan with intravenous or oral contrast if the contrast is not medically contraindicated or MRI
  * Brain: CT scan or MRI
  * Bone: Whole body Bone Scintigraphy
* Patients must meet the following laboratory criteria within 2 weeks (14 days) prior to registration:
* Hematology
* Neutrophil count of > 1200/mm3
* Platelet count of > 100,000/mm3
* Hemoglobin ≥ 90 g/L
* Biochemistry
* AST/SGOT and ALT/SGPT ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if the transaminase elevation is due to disease involvement
* Serum bilirubin ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 50 mL/min
* Serum potassium, sodium, magnesium, phosphorus, and calcium within normal limits for the institution
* Serum albumin ≥ LLN or 30g/L
* Clinically euthyroid function (TSH and free T4). (Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism).
* LVEF assessment (2-D echocardiogram or MUGA scan) performed within 6 weeks prior to registration, showing a LVEF value > 50%
* Electrocardiogram performed within 1 week prior to registration (details about findings on the Electrocardiogram that are not acceptable for participating in the study are reported in the Exclusion criteria section)
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to registration and agree to appropriate method of pregnancy prevention.
* Patient should have an archival tumor sample available for confirmation of HER2, Estrogen and Progesterone status by the central lab.

Exclusion Criteria:

* Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
* Patients who need valproic acid for any other medical condition during the study or within 5 days prior to first panobinostat treatment
* Patients who have received prior systemic anti-cancer therapy (cytotoxic chemotherapy, endocrine therapy, targeted therapy, monoclonal antibody or biologic therapy) or investigational agent within the last 4 weeks prior to registration (6 weeks for nitrosoureas and mitomycin; 2 weeks for capecitabine)
* Patients who have received prior radiotherapy to ≥ 25% of the bone marrow within the last 4 weeks prior to registration; local radiotherapy is allowed however all recently irradiated lesions should not be included in the measurable disease assessment.
* Patients who have received prior investigational agents within the last 4 weeks prior to registration
* Patients with unresolved diarrhea ≥CTCAE grade 1
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral panobinostat
* History of cardiac dysfunction including any one of the following:
* Complete left bundle branch block or obligate use of a cardiac pacemaker or congenital long QT syndrome or history or presence of ventricular tachyarrhythmias or clinically significant resting bradycardia (<50 beats per minute) or QTcF > 450 msec on screening ECG or right bundle branch block and left anterior hemiblock (bifascicular block)
* Presence of unstable atrial fibrillation (ventricular response rate >100 bpm). Patients with stable atrial fibrillation are allowed in the study provided they do not meet the other cardiac exclusion criteria
* Previous history angina pectoris or acute MI within 6 months of registration
* Congestive Heart Failure (New York Heart Association functional classification III-IV)
* History of unexplained syncope
* Other clinically significant heart disease (e.g. cardiomyopathy, cardiac artery disease, uncontrolled hypertension, or history of poor compliance with an antihypertensive regimen)
* Family history of long QT syndrome, unexplained syncope or unexplained sudden death
* Acute or chronic liver or renal disease
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes mellitus, active untreated or uncontrolled infection, chronic obstructive or chronic restrictive pulmonary disease including dyspnoea at rest from any cause) that could cause unacceptable safety risks or compromise compliance with the protocol
* Concomitant use of drugs with a risk of causing torsades de pointes where such treatments cannot be discontinued or switched to a different medication prior to starting study drug
* Brain metastases, unless patient randomized on study at least 90 days from completion of brain radiotherapy and / or surgery without radiologic or functional evidence of progressive brain metastases, and off corticosteroids above the dose of 7.5 mg prednisone or equivalent; No concurrent radiotherapy for brain metastasis is allowed
* Clinically significant third space fluid accumulation
* Concurrent biphosphonates unless if initiated prior to study entry (at least 4 weeks before patient registration)
* Pregnant (i.e., positive beta-human chorionic gonadotropin test) or breast feeding patient
* Unable to swallow oral medications
* Not willing to use a double barrier method of non-hormonal birth control. Contraception must be used during the study and for 30 days after last dose of study treatment.
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hurvitz, MD, Study Chair — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ER+ and/or PgR+ (Arm I); ER- and PgR- (Arm II): Panobinostat - LBH589: hard gelatine capsule - 5mg and 20mg
Period: Overall Study
Arm/Group | ER+ and/or PgR+ (Arm I) | ER- and PgR- (Arm II)
Started | 33 | 21
Completed | 32 | 20
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — No treatment (elevated liver enzymes) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ER+ and/or PgR+ (Arm I) | ER- and PgR- (Arm II) | Total
Number analyzed (Participants) | 33 | 21 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 18 | 40
  >=65 years | 11 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (9.5) | 52.8 (10.7) | 57.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 21 | 54
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Race - White | 31 | 20 | 51
  Race - Black or African American | 1 | 0 | 1
  Race - Asian | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21
  Belgium | 1 | 0 | 1
  Canada | 4 | 6 | 10
  France | 5 | 1 | 6
  Ireland | 10 | 1 | 11
  United Kingdom | 2 | 3 | 5
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 31 | 18 | 49
Menopausal Status [Number; unit: participants]
  Premenopausal | 0 | 5 | 5
  Postmenopausal | 33 | 16 | 49

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (as Determined by Investigator): the Percentage of Patients Assigned to a Treatment Arm With a Confirmed Best Response of CR or PR.
Description: The assessment of overall response (OR) is based on the response of target lesion, of non-target lesion, and on presence of new lesions (RECIST criteria version 1.0 using imaging techniques; as per investigator assessment).
Time Frame: 6 years and 2 months
Measure: Number; unit: participants
Arm/Group | ER+ and/or PgR+ (Arm I) | ER- and PgR- (Arm II)
Number analyzed (Participants) | 33 | 21
participants
  Complete Response | 0 | 1
  Partial Response | 1 | 0
  Stable Disease / Incompete Response | 13 | 4
  Progressive Disease | 14 | 14
  Missing | 5 | 2

ADVERSE EVENTS:
Description: Patients were regularly evaluated for AEs at each study visit, and carefully monitored during the entire treatment phase. Safety evaluations consisted of medical interviews, recording of AEs as reported by the patient, physical examinations, blood pressure, and laboratory measurements.
Arm/Group | ER+ and/or PgR+ (Arm I) | ER- and PgR- (Arm II)
Serious Adverse Events (participants affected / at risk) | 12/32 | 8/20
Other Adverse Events (participants affected / at risk) | 32/32 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ER+ and/or PgR+ (Arm I) (N=32) | ER- and PgR- (Arm II) (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ER+ and/or PgR+ (Arm I) (N=32) | ER- and PgR- (Arm II) (N=20)
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 4
Palpitations (Cardiac disorders) | 0 | 3
Hyperthyroidism (Endocrine disorders) | 3 | 1
Lacrimation increased (Eye disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 12 | 5
Diarrhoea (Gastrointestinal disorders) | 25 | 15
Dry mounth (Gastrointestinal disorders) | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Haemorrhoids (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 28 | 16
Stomatitis (Gastrointestinal disorders) | 6 | 1
Vomiting (Gastrointestinal disorders) | 24 | 11
Asthenia (General disorders) | 1 | 2
Chest pain (General disorders) | 1 | 3
Fatigue (General disorders) | 26 | 15
Mucosal inflammation (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 3
Oedema (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 5 | 7
Pain (General disorders) | 1 | 5
Pyrexia (General disorders) | 2 | 2
Infection (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Oral herpes (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Upper respiratory infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Electrocardiogram abnormal (Investigations) | 2 | 0
Weight decreased (Investigations) | 8 | 2
Decreased appetite (Metabolism and nutrition disorders) | 14 | 10
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 5
Dizziness (Nervous system disorders) | 5 | 3
Dysgeusia (Nervous system disorders) | 8 | 4
Headache (Nervous system disorders) | 5 | 5
Lethargy (Nervous system disorders) | 0 | 3
Neuralgia (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 5 | 3
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2

LIMITATIONS AND CAVEATS:
In Arm II, low recruitment resulted in insufficient data (and enrollment was stopped). In Arm I, the required number of tumor responses was not reached. Unable to determine efficacy (small sample); secondary objectives also removed from the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No